CLINICAL TRIAL: NCT02342808
Title: Treating Resistant Hypertension Using Lifestyle Modification to Promote Health
Brief Title: Lifestyle Interventions in Treatment-Resistant Hypertension
Acronym: TRIUMPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Pro00055703; 1R01HL122836-01A1 (NIH)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Treatment-Resistant Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structured center-based lifestyle intervention (Experimental): The Structured center-based Lifestyle Intervention (C-LIFE) will include individualized plans for the DASH diet, weight management, and aerobic exercise.
  Interventions: Behavioral: Structured center-based lifestyle intervention
- Standard education and physician advice (Experimental): The Medical Management with Standardized Education and Physician Advice (SEPA) will consist of encouragement to achieve an ideal body weight and engage in exercise as part of routine counseling in primary care, but no special program will be delivered to enhance the participants' ability to comply with these recommendations.
  Interventions: Behavioral: Standard education and physician advice

INTERVENTIONS:
Behavioral: Structured center-based lifestyle intervention — Participants will meet with interventionists weekly for 16 weeks and receive instruction on the DASH diet with caloric and sodium restriction and will exercise three times per week at one of the designated CR facilities, under the supervision of medically trained staff, 3 times per week for 16 weeks.
  Arms: Structured center-based lifestyle intervention
Behavioral: Standard education and physician advice — Participants will receive routine medical care provided by the participants' primary care physician(s) supplemented by an educational session on hypertension management. Participants will receive a dietary consultation from the study nutritionist and an individualized exercise prescription from an exercise physiologist, but not participate in a structured program. Participants will be free to engage in diet and exercise for the 16-week intervention.
  Arms: Standard education and physician advice

SUMMARY:
This study will examine the effects of lifestyle intervention on fitness, dietary habits, and body weight in patients with resistant hypertension (RH). Patients will be randomized to either a 4-month adjunctive lifestyle intervention designed to lower BP that will be delivered in a center-based CR program (C-LIFE), or to standardized education and physician advice (SEPA) designed to promote the same healthy behaviors and reflecting the current highest possible standard of care for promoting a healthy lifestyle in RH.

DETAILED DESCRIPTION:
The term resistant hypertension (RH) is defined as clinic blood pressure (BP) that remains above goal (e.g., systolic blood pressure [SBP]>140 mm Hg and/or diastolic blood pressure [DBP]>90 mm Hg), despite adherence to a regimen of 3 or more antihypertensive medications of different classes, one of which is a diuretic.

With the growing prevalence of hypertension (HTN) in this country, RH is a major public health concern, affecting more than 7.5 million Americans. Patients with RH are 50% more likely to experience a CVD event, including stroke, kidney failure, myocardial infarction, and death, compared to patients with controlled BP. There is an urgent need for developing RH management strategies to lower BP as well as to reduce the high risk of CVD-related events. Lifestyle modifications, including exercise training and dietary modification, are of proven efficacy in lowering BP in unmedicated patients with HTN and are often recommended as the first step for treating high BP. The Dietary Approaches to Stop Hypertension (DASH) diet has been shown to lower BP in HTN patients who are not treated with drugs. Moreover, when the DASH diet is combined with exercise and caloric restriction, even greater, and quite marked, BP reductions can be achieved. However, the efficacy of these lifestyle modifications in HTN patients who are refractory to medical therapy is unknown. This application aims to build upon evidence supporting the value of lifestyle modifications in unmedicated patients with HTN by proposing a randomized clinical trial (RCT) that will evaluate whether an intensive, medically-supervised lifestyle intervention can successfully lower BP in medicated patients with RH.

ELIGIBILITY:
Inclusion Criteria:

* Documented resistant hypertension (RH). In the absence of a specific RH diagnosis, individuals being treated for two or more weeks with 3 antihypertensive medications of different classes, including a diuretic if tolerated, with clinic SBP ≥ 130 mm Hg or DBP ≥ 80 mm Hg, will be eligible. Individuals being treated with 4 or more antihypertensive medications, including a diuretic if tolerated, with SBP ≥ 120 or DBP ≥ 80 mm Hg will also be eligible.
* Adherent to prescribed medications
* Overweight (BMI ≥ 25 kg/m2)
* Sedentary
* Willing to be randomized to one of the 2 treatment groups and able to fully participate in intervention
* Informed consent

Exclusion Criteria:

* Secondary HTN, non-adherence to anti-HTN medications
* Severe CKD (eGFR <40 ml/min/1.73m2)
* Severe ischemic heart disease (CCS Class 3 or 4 angina or evidence of ischemia at <85% heart rate reserve on treadmill testing)
* Severe heart failure (NYHA association Class 3 or 4), high grade arrhythmias, severe valvular heart disease
* Severe asthma or chronic obstructive lung disease
* Diabetes requiring insulin
* Musculoskeletal or neurologic problems that would preclude participation in aerobic exercise training
* Major psychiatric disorder, a history of drug abuse, alcohol consumption >14 drinks/week
* Life-limiting comorbid medical condition such as cancer
* Prior gastric bypass surgery
* Currently pregnant
* Cognitively impaired

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-06; Primary Completion 2020-05-08 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Change in clinic systolic blood pressure | Baseline to immediate post-treatment (4 months)

SECONDARY OUTCOMES:
Change in 24-hour ambulatory systolic blood pressure | Baseline to immediate post-treatment (4 months)
Weight | Immediate post-treatment (4 months)
Aerobic capacity (Measured via an exercise treadmill stress test with VO2 collection) | Immediate post-treatment (4 months)
  Measured via an exercise treadmill stress test with VO2 collection
DASH Diet adherence (Measured via food diary recall) | Immediate post-treatment (4 months)
  Measured via food diary recall
Change in Cardiovascular Disease (CVD) biomarker composite score | Baseline to immediate post-treatment (4 months)
  Biomarkers of interest include: left ventricular hypertrophy, arterial stiffness, baroreceptor reflex sensitivity, insulin resistance, lipid profiles, sympathetic nervous system (SNS) activity, and inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: James A. Blumenthal, PhD, Principal Investigator — Duke University; Andrew Sherwood, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Blumenthal JA, Smith PJ, Mabe S, Hinderliter A, Craighead L, Watkins LL, Ingle K, Tyson CC, Lin PH, Kraus WE, Liao L, Sherwood A. Effects of Lifestyle Modification on Psychosocial Function in Patients With Resistant Hypertension: SECONDARY OUTCOMES FROM THE TRIUMPH RANDOMIZED CLINICAL TRIAL. J Cardiopulm Rehabil Prev. 2024 Jan 1;44(1):64-70. doi: 10.1097/HCR.0000000000000801. Epub 2023 May 24. PMID 37220236
- [Derived] Blumenthal JA, Hinderliter AL, Smith PJ, Mabe S, Watkins LL, Craighead L, Ingle K, Tyson C, Lin PH, Kraus WE, Liao L, Sherwood A. Effects of Lifestyle Modification on Patients With Resistant Hypertension: Results of the TRIUMPH Randomized Clinical Trial. Circulation. 2021 Oct 12;144(15):1212-1226. doi: 10.1161/CIRCULATIONAHA.121.055329. Epub 2021 Sep 27. PMID 34565172
- [Derived] Smith PJ, Mabe SM, Sherwood A, Doraiswamy PM, Welsh-Bohmer KA, Burke JR, Kraus WE, Lin PH, Browndyke JN, Babyak MA, Hinderliter AL, Blumenthal JA. Metabolic and Neurocognitive Changes Following Lifestyle Modification: Examination of Biomarkers from the ENLIGHTEN Randomized Clinical Trial. J Alzheimers Dis. 2020;77(4):1793-1803. doi: 10.3233/JAD-200374. PMID 32925039
- [Derived] Blumenthal JA, Sherwood A, Smith PJ, Mabe S, Watkins L, Lin PH, Craighead LW, Babyak M, Tyson C, Young K, Ashworth M, Kraus W, Liao L, Hinderliter A. Lifestyle modification for resistant hypertension: The TRIUMPH randomized clinical trial. Am Heart J. 2015 Nov;170(5):986-994.e5. doi: 10.1016/j.ahj.2015.08.006. Epub 2015 Aug 14. PMID 26542509